CLINICAL TRIAL: NCT03482804
Title: The Inclined Position in Case of Respiratory Discomfort in the One Year Less Infant : Study on the Profits and the Risks in the Home
Acronym: PROCLIVE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0161
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Obstruction, Airway; Sudden; Death, Infant
MeSH Terms: conditions — Airway Obstruction; Sudden Infant Death | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — Parents will be interviewed before being seen in consultation in the emergency room. The reason for consultation will not be taken into account, the only criterion being the age of the child. There will be no sign in the waiting room, the study will be proposed to them by the principal investigator.
  The questionnaires will be collected on live paper. The answers will be transferred in a second time on an Excel database protected by a password.

SUMMARY:
The inclined position at 30 ° in case of transient respiratory discomfort is recommended since the consensus conference of September 2000. This recommendation is based on a low level of evidence (grade C). This advice is found in the health book, and in many tips for parents. However, it does not comply with the recommendations of the American Academy of Pediatrics for sleeping on the back, on a firm mattress and without other objects in the bed.

70% of pediatricians advise this position in a specific medical context according to a study of Bellaïche conducted in 2013. 40% of parents use it for no particular reason.

Anatomically, the upper airways of infants are of reduced caliber, and therefore at risk of obstruction.

A study by Bergougnioux on the cases of MIN in infants wearing a wrap-around sling shows that the flexion of the neck causes the chin to be positioned against the chest and contributes to the suffocation of the infant. This is especially important in infants under 3 months whose neck muscles do not yet support the weight of the head.

The 2009 InVS national survey of unexpected infant deaths shows that bed crashes accounted for 11.1% of all deaths reported. Among unexplained deaths, maladaptive bedding was a contributing factor, including the use of a pillow in the bed in 24.3% of cases.

It was observed in the study by Kornhauser Cerar et al in 2009 that half-sitting in a car seat for an extended duration was at the origin of a significant desaturations rate, which was also found in the car bed group. The control group "hospital bed" was not subject to these desaturations. These results support the fact that only an adapted bedding that complies with the recommendations protects against asphyxiation.

Since 2016, INPES recommends in its advice sheet on bronchiolitis for parents, a flat bed on the back.

Hypothesis :

The inclined position in infants under one year of age is at risk of unexpected death of the infant by obstruction of the upper airways, because of the changes of position that it entails, including a risk of slipping at the bottom of the bed and of asphyxiation under the covers.

ELIGIBILITY:
Inclusion Criteria:

* Infant from 0 to 12 months
* Lie in a proclive position while sleeping
* Whose parents / parent authority holders informed about the terms of the study and agree to answer the questionnaire

Exclusion Criteria:

* Refusal to participate

Max Age: 12 Months | Sex: All
Age Groups: Child
Study Population: Parents of infants from 0 to 12 months attending pediatric emergencies in 2 hospitals are interroged :
  * Hôpital Femme Mere Enfant (Bron)
  * Hôpital Nord-Ouest (Villefranche sur Saône) Are included infant from 0 to 12 months, lie in a proclive position while sleeping whose parents / parent authority holders informed about the terms of the study and agree to answer the questionnaire
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Sliding of the infant in the bottom of his bed in inclined position during sleep | 1 day
  Sliding of the infant in the bottom of his bed in inclined position during sleep, reported by the parents during the questionnaire in the form of a closed question.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Femme Mère Enfant, Bron
  - Accueil des urgences pédiatriques - Hôpital Nord-Ouest Villefranche sur Saône, Gleizé

IPD SHARING:
Plan to Share IPD: No